CLINICAL TRIAL: NCT00300430
Title: A Long-Term, Open-Label, Safety Extension Study of the Combination of Fenofibric Acid and Statin Therapy for Subjects With Mixed Dyslipidemia
Brief Title: Study to Evaluate the Long-Term Safety and Efficacy of ABT-335, in Combination With Three Different Statins in Subjects With Mixed Dyslipidemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Maureen Kelly, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M05-758
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-06

CONDITIONS: Dyslipidemia; Coronary Heart Disease; Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Coronary Disease | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium; Fenofibrate; Atorvastatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): 20 mg drug and ABT-335
  Interventions: Drug: ABT-335 and rosuvastatin calcium
- B (Active Comparator): 40 mg drug and ABT 335
  Interventions: Drug: ABT-335 and atorvastatin calcium
- C (Active Comparator): 40 mg drug and ABT-335
  Interventions: Drug: ABT-335 and simvastatin

INTERVENTIONS:
Drug: ABT-335 and rosuvastatin calcium — ABT-335 135 mg plus rosuvastatin calcium daily, 52 weeks
  Other Names: ABT-335; TRILIPIX
  Arms: A
Drug: ABT-335 and atorvastatin calcium — ABT-335 135 mg plus atorvastatin calcium daily, 52 weeks
  Other Names: ABT-335; TRILIPIX
  Arms: B
Drug: ABT-335 and simvastatin — ABT-335 135 mg plus simvastatin daily, 52 weeks
  Other Names: ABT-335; TRILIPIX
  Arms: C

SUMMARY:
The primary purpose of this study is to test the safety and the effects of using an investigational drug regimen; once daily ABT-335 (Investigational drug) administered in combination with once daily atorvastatin calcium, rosuvastatin calcium or simvastatin in patients with abnormal lipid levels in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects who voluntarily sign the informed consent.
* Subject has successfully completed one of the three ABT-335, rosuvastatin, simvastatin and atorvastatin combination therapy studies.

Exclusion Criteria:

* Subject is using or will use investigational medications, except as approved by Abbott.
* Subject has prematurely discontinued his/her initial therapy one of the prior ABT-335, rosuvastatin, simvastatin and atorvastatin calcium combination therapy studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1911 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Global Medical Information, North Chicago, Illinois, United States

REFERENCES:
- [Derived] Ferdinand KC, Davidson MH, Kelly MT, Setze CM. One-year efficacy and safety of rosuvastatin + fenofibric acid combination therapy in patients with mixed dyslipidemia: evaluation of dose response. Am J Cardiovasc Drugs. 2012 Apr 1;12(2):117-25. doi: 10.2165/11597940-000000000-00000. PMID 22263674
- [Derived] Jones PH, Bays HE, Davidson MH, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Evaluation of a new formulation of fenofibric acid, ABT-335, co-administered with statins : study design and rationale of a phase III clinical programme. Clin Drug Investig. 2008;28(10):625-34. doi: 10.2165/00044011-200828100-00003. PMID 18783301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1895 subjects were treated in this study. 306 others who did not enroll in this study but were treated with combo therapy in preceding double-blind studies are included in analyses of adverse events. Six subjects were enrolled, but never received study drug. An additional 10 subjects from a site that was closed were not included in any analysis.
Groups:
- ABT-335 + 20 mg Rosuvastatin: ABT-335 and 20 mg rosuvastatin combination therapy
- ABT-335 + 40 mg Simvastatin: ABT-335 and 40 mg simvastatin combination therapy
- ABT-335 + 40 mg Atorvastatin: ABT-335 and 40 mg atorvastatin combination therapy
Period: Overall Study
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Started | 1186 ("Started" = received combo therapy in double-blind and/or open-label study.) | 514 ("Started" = received combo therapy in double-blind and/or open-label study.) | 501 ("Started" = received combo therapy in double-blind and/or open-label study.)
Completed | 819 ("Completed" = completed both the double-blind and open-label studies.) | 345 ("Completed" = completed both the double-blind and open-label studies.) | 350 ("Completed" = completed both the double-blind and open-label studies.)
Not Completed | 367 | 169 | 151

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin | Total
Number analyzed (Participants) | 1186 | 514 | 501 | 2201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 965 | 440 | 397 | 1802
  >=65 years | 221 | 74 | 103 | 398
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.79) | 54.1 (10.25) | 55.5 (10.86) | 55.0 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 608 | 256 | 256 | 1120
  Male | 578 | 258 | 245 | 1081
Region of Enrollment [Number; unit: participants]
  North America | 1186 | 514 | 501 | 2201

OUTCOME MEASURES:

1. Secondary Outcome: Median Percent Change in Triglycerides From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: Subjects who took at least 1 dose of ABT-335 plus a statin in the preceding double-blind studies. Baseline is the last value before the first dose of combination therapy in the preceding studies. Percent changes from baseline to Week 52 in this open-label study are summarized. No imputations were made for missing values.
Measure: Median (Full Range); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 284 | 120 | 122
percent change | -53.0 (27.67) [-92.7 to 87.9] | -47.7 (24.62) [-89.7 to 74.8] | -56.2 (24.56) [-92.5 to 60.7]

2. Secondary Outcome: Mean Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 284 | 120 | 121
percent change | 25.2 (23.22) | 25.1 (25.08) | 19.4 (20.58)

3. Secondary Outcome: Mean Percent Change in Direct Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 283 | 120 | 121
percent change | -41.6 (20.77) | -30.2 (21.83) | -38.1 (19.09)

4. Secondary Outcome: Mean Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 52 in This Open-label Study
Time Frame: Baseline to Week 52 in this open-label study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 284 | 120 | 121
percent change | -48.8 (15.80) | -36.6 (16.90) | -44.3 (15.72)

5. Secondary Outcome: Mean Percent Change in Very Low-density Lipoprotein Cholesterol (VLDL-C) From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 272 | 117 | 122
percent change | -56.9 (27.85) | -37.7 (63.12) | -52.2 (36.54)

6. Secondary Outcome: Mean Percent Change in Total Cholesterol From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 284 | 120 | 122
percent change | -37.9 (13.14) | -27.5 (14.60) | -35.0 (13.01)

7. Secondary Outcome: Mean Percent Change in Apolipoprotein B (Apo B) From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 277 | 115 | 120
percent change | -44.8 (15.40) | -35.5 (14.85) | -42.9 (14.23)

8. Primary Outcome: Percentage of Subjects Reporting Adverse Events During Combination Therapy, Either in the Preceding Double-blind Studies or in This Open-label Study
Time Frame: Anytime after initiation of combination therapy (either in the double-blind or open-label study) to within 30 days after the last dose of combination therapy
Population: Subjects who took at least 1 dose of ABT-335 plus a statin in the preceding double-blind studies or in this open-label study. All adverse events in the preceding studies or in this study occurring with exposure to combination therapy are summarized.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 1186 | 514 | 501
percentage of participants | 83 | 86 | 85

9. Secondary Outcome: Median Percent Change in High-sensitivity C-reactive Protein (hsCRP) From Baseline to Week 52 of the Open-label Study
Time Frame: Baseline to Week 52 of the open-label study
Population: as for outcome 1
Measure: Median (Full Range); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 279 | 117 | 120
percent change | -38.87 (265.37) [-94.5 to 1166.0] | -27.72 (93.62) [-99.8 to 2558.5] | -39.13 (70.99) [-95.4 to 384.3]

ADVERSE EVENTS:
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Serious Adverse Events (participants affected / at risk) | 85 | 40 | 23
Other Adverse Events (participants affected / at risk) | 646 | 308 | 283
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Anemia (Blood and lymphatic system disorders) | 1/1186 | 0/514 | 0/501
Acute coronary syndrome (Cardiac disorders) | 0/1186 | 1/514 | 0/501
Acute myocardial infarction (Cardiac disorders) | 1/1186 | 1/514 | 0/501
Angina pectoris (Cardiac disorders) | 1/1186 | 1/514 | 0/501
Angina unstable (Cardiac disorders) | 0/1186 | 0/514 | 1/501
Atrial fibrillation (Cardiac disorders) | 0/1186 | 1/514 | 0/501
Atrial flutter (Cardiac disorders) | 2/1186 | 1/514 | 0/501
Cardiac arrest (Cardiac disorders) | 0/1186 | 1/514 | 0/501
Cardiac failure congestive (Cardiac disorders) | 1/1186 | 0/514 | 0/501
Cardio-respiratory arrest (Cardiac disorders) | 0/1186 | 0/514 | 1/501
Coronary artery disease (Cardiac disorders) | 5/1186 | 0/514 | 0/501
Mitral valve incompetence (Cardiac disorders) | 0/1186 | 1/514 | 0/501
Myocardial infarction (Cardiac disorders) | 4/1186 | 1/514 | 0/501
Myocardial ischemia (Cardiac disorders) | 1/1186 | 0/514 | 0/501
Pericarditis (Cardiac disorders) | 1/1186 | 0/514 | 0/501
Sick sinus syndrome (Cardiac disorders) | 0/1186 | 1/514 | 0/501
Ventricular tachycardia (Cardiac disorders) | 0/1186 | 1/514 | 0/501
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1/1186 | 0/514 | 0/501
Hyperparathyroidism primary (Endocrine disorders) | 1/1186 | 0/514 | 0/501
Retinal detachment (Eye disorders) | 0/1186 | 1/514 | 0/501
Vitreous detachment (Eye disorders) | 1/1186 | 0/514 | 0/501
Abdominal hernia (Gastrointestinal disorders) | 0/1186 | 1/514 | 0/501
Abdominal pain upper (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Duodenitis (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Dysphagia (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Enterocele (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0/1186 | 1/514 | 0/501
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Nausea (Gastrointestinal disorders) | 0/1186 | 0/514 | 1/501
Pancreatitis (Gastrointestinal disorders) | 1/1186 | 0/514 | 1/501
Pancreatitis acute (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Small intestinal obstruction (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Umbilical hernia (Gastrointestinal disorders) | 0/1186 | 2/514 | 0/501
Vomiting (Gastrointestinal disorders) | 1/1186 | 0/514 | 0/501
Chest discomfort (General disorders) | 1/1186 | 0/514 | 2/501
Chest pain (General disorders) | 2/1186 | 1/514 | 2/501
Non-cardiac chest pain (General disorders) | 1/1186 | 1/514 | 0/501
Bile duct obstruction (Hepatobiliary disorders) | 0/1186 | 1/514 | 0/501
Cholecystitis (Hepatobiliary disorders) | 2/1186 | 0/514 | 1/501
Cholecystitis acute (Hepatobiliary disorders) | 2/1186 | 0/514 | 0/501
Cholecystitis chronic (Hepatobiliary disorders) | 0/1186 | 1/514 | 0/501
Cholelithiasis (Hepatobiliary disorders) | 0/1186 | 1/514 | 1/501
Latex allergy (Immune system disorders) | 0/1186 | 1/514 | 0/501
Abdominal wall infection (Infections and infestations) | 0/1186 | 1/514 | 0/501
Appendicitis (Infections and infestations) | 0/1186 | 1/514 | 0/501
Bacteremia (Infections and infestations) | 1/1186 | 0/514 | 0/501
Cellulitis (Infections and infestations) | 1/1186 | 0/514 | 0/501
Diverticulitis (Infections and infestations) | 4/1186 | 0/514 | 0/501
Gastroenteritis (Infections and infestations) | 1/1186 | 0/514 | 0/501
Gastroenteritis viral (Infections and infestations) | 1/1186 | 0/514 | 0/501
Hepatitis viral (Infections and infestations) | 0/1186 | 0/514 | 1/501
Orchitis (Infections and infestations) | 0/1186 | 1/514 | 0/501
Pneumonia (Infections and infestations) | 1/1186 | 1/514 | 0/501
Pneumonia pneumococcal (Infections and infestations) | 1/1186 | 0/514 | 0/501
Postoperative wound infection (Infections and infestations) | 1/1186 | 0/514 | 0/501
Subcutaneous abscess (Infections and infestations) | 1/1186 | 0/514 | 0/501
Upper respiratory tract infection (Infections and infestations) | 1/1186 | 0/514 | 0/501
Urinary tract infection (Infections and infestations) | 1/1186 | 0/514 | 0/501
Accidental overdose (Injury, poisoning and procedural complications) | 1/1186 | 0/514 | 1/501
Device failure (Injury, poisoning and procedural complications) | 0/1186 | 0/514 | 1/501
Hip fracture (Injury, poisoning and procedural complications) | 0/1186 | 0/514 | 1/501
Humerus fracture (Injury, poisoning and procedural complications) | 1/1186 | 0/514 | 0/501
Incisional hernia (Injury, poisoning and procedural complications) | 1/1186 | 0/514 | 0/501
Limb injury (Injury, poisoning and procedural complications) | 0/1186 | 1/514 | 0/501
Post procedural hematoma (Injury, poisoning and procedural complications) | 0/1186 | 1/514 | 0/501
Post procedural sepsis (Injury, poisoning and procedural complications) | 1/1186 | 0/514 | 0/501
Postoperative fever (Injury, poisoning and procedural complications) | 1/1186 | 0/514 | 0/501
Skin laceration (Injury, poisoning and procedural complications) | 0/1186 | 1/514 | 0/501
Blood pressure increased (Investigations) | 0/1186 | 0/514 | 1/501
Ultrasound kidney abnormal (Investigations) | 0/1186 | 0/514 | 1/501
Obesity (Metabolism and nutrition disorders) | 1/1186 | 0/514 | 0/501
Back pain (Musculoskeletal and connective tissue disorders) | 1/1186 | 1/514 | 0/501
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/1186 | 0/514 | 0/501
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1/1186 | 0/514 | 0/501
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3/1186 | 1/514 | 0/501
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/1186 | 0/514 | 0/501
Neck pain (Musculoskeletal and connective tissue disorders) | 1/1186 | 0/514 | 0/501
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6/1186 | 4/514 | 0/501
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1/1186 | 0/514 | 0/501
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/1186 | 0/514 | 0/501
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/1186 | 1/514 | 0/501
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Carcinoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 1/514 | 0/501
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1186 | 0/514 | 1/501
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1186 | 0/514 | 1/501
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1186 | 0/514 | 0/501
Brain edema (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Brain stem infarction (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Carotid artery stenosis (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Cerebrovascular accident (Nervous system disorders) | 0/1186 | 1/514 | 1/501
Dementia (Nervous system disorders) | 0/1186 | 1/514 | 0/501
Dizziness (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Dysarthria (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Grand mal convulsion (Nervous system disorders) | 0/1186 | 1/514 | 0/501
Headache (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Hydrocephalus (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Lethargy (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Migraine (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Normal pressure hydrocephalus (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Presyncope (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Somnolence (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Syncope (Nervous system disorders) | 2/1186 | 1/514 | 1/501
Transient ischemic attack (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Trigeminal neuralgia (Nervous system disorders) | 0/1186 | 0/514 | 1/501
Unresponsive to stimuli (Nervous system disorders) | 1/1186 | 0/514 | 0/501
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/1186 | 1/514 | 1/501
Anxiety disorder (Psychiatric disorders) | 1/1186 | 1/514 | 0/501
Confusional state (Psychiatric disorders) | 1/1186 | 0/514 | 0/501
Major depression (Psychiatric disorders) | 0/1186 | 1/514 | 0/501
Mental status changes (Psychiatric disorders) | 1/1186 | 0/514 | 0/501
Calculus ureteric (Renal and urinary disorders) | 1/1186 | 0/514 | 0/501
Glomerulonephritis proliferative (Renal and urinary disorders) | 1/1186 | 0/514 | 0/501
Hematuria (Renal and urinary disorders) | 1/1186 | 0/514 | 0/501
Nephrolithiasis (Renal and urinary disorders) | 0/1186 | 1/514 | 0/501
Renal colic (Renal and urinary disorders) | 1/1186 | 0/514 | 1/501
Renal failure acute (Renal and urinary disorders) | 0/1186 | 1/514 | 0/501
Renal impairment (Renal and urinary disorders) | 0/1186 | 1/514 | 0/501
Cystocele (Reproductive system and breast disorders) | 1/1186 | 0/514 | 0/501
Menorrhagia (Reproductive system and breast disorders) | 1/1186 | 0/514 | 0/501
Menstruation irregular (Reproductive system and breast disorders) | 1/1186 | 0/514 | 0/501
Ovarian cyst (Reproductive system and breast disorders) | 1/1186 | 0/514 | 0/501
Rectocele (Reproductive system and breast disorders) | 1/1186 | 0/514 | 0/501
Uterine pain (Reproductive system and breast disorders) | 1/1186 | 0/514 | 0/501
Uterine prolapse (Reproductive system and breast disorders) | 2/1186 | 0/514 | 1/501
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/1186 | 0/514 | 0/501
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/1186 | 0/514 | 0/501
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/1186 | 0/514 | 0/501
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/1186 | 0/514 | 1/501
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0/1186 | 1/514 | 0/501
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/1186 | 0/514 | 0/501
Aortic aneurysm (Vascular disorders) | 0/1186 | 1/514 | 0/501
Deep vein thrombosis (Vascular disorders) | 4/1186 | 1/514 | 1/501
Femoral arterial stenosis (Vascular disorders) | 0/1186 | 0/514 | 1/501
Hypotension (Vascular disorders) | 1/1186 | 0/514 | 1/501
Intermittent claudication (Vascular disorders) | 1/1186 | 0/514 | 0/501
Thrombophlebitis superficial (Vascular disorders) | 1/1186 | 0/514 | 0/501
Thrombosis (Vascular disorders) | 0/1186 | 0/514 | 1/501
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Diarrhea (Gastrointestinal disorders) | 49/1186 | 26/514 | 33/501
Dyspepsia (Gastrointestinal disorders) | 42/1186 | 31/514 | 28/501
Nausea (Gastrointestinal disorders) | 61/1186 | 23/514 | 34/501
Bronchitis (Infections and infestations) | 60/1186 | 25/514 | 23/501
Nasopharyngitis (Infections and infestations) | 116/1186 | 70/514 | 58/501
Sinusitis (Infections and infestations) | 91/1186 | 40/514 | 37/501
Upper respiratory tract infection (Infections and infestations) | 145/1186 | 69/514 | 57/501
Arthralgia (Musculoskeletal and connective tissue disorders) | 86/1186 | 54/514 | 38/501
Back pain (Musculoskeletal and connective tissue disorders) | 118/1186 | 56/514 | 42/501
Muscle spasms (Musculoskeletal and connective tissue disorders) | 55/1186 | 34/514 | 35/501
Myalgia (Musculoskeletal and connective tissue disorders) | 60/1186 | 27/514 | 25/501
Pain in extremity (Musculoskeletal and connective tissue disorders) | 53/1186 | 32/514 | 33/501
Headache (Nervous system disorders) | 160/1186 | 75/514 | 74/501
Cough (Respiratory, thoracic and mediastinal disorders) | 49/1186 | 35/514 | 32/501
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 23/1186 | 26/514 | 21/501

LIMITATIONS AND CAVEATS:
This was an open-label study designed to assess the longer-term safety of the combination therapies. Evaluation of efficacy outcomes was a secondary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not to publish or present the results before the publication of the multi-center investigator paper, but in no event shall be so restricted after the expiration of twelve (12) months from completion of the studies at all sites. Any presentation or publication to be submitted to Sponsor (in draft of the same) for Sponsor review and comment.